CLINICAL TRIAL: NCT06919419
Title: The HOTSPOT Study Hybrid Implementation-effectiveness Study to Optimize HIV Testing and PrEP in a Southern Jail
Brief Title: HOTSPOT Study: Implement and Evaluate the PrEP (Pre-exposure Prophylaxis) Implementation Strategy
Acronym: Hotspot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ank Nijhawan, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STU-2024-1096; 1R01MH129185-01 (NIH)
Record Dates: First submitted 2025-03-21; First posted 2025-04-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: PrEP; HIV; Incarceration

STUDY DESIGN:
Intervention Model Description: Patients identified to be at elevated risk for HIV will meet with the PrEP navigator during incarceration
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PrEP navigation (Other): This is a single arm study where people in the Dallas County Jail identified to be at elevated risk for HIV are offered a PrEP navigation visit
  Interventions: Behavioral: Multicomponent strategy

INTERVENTIONS:
Behavioral: Multicomponent strategy — Identify patients for HIV/STI testing, engage in discussions around PrEP and navigate patients to PrEP after jail incarceration

SUMMARY:
The goal of this study is to measure the implementation and effectiveness of a multicomponent strategy for PrEP for people who are incarcerated at the Dallas County Jail. Specifically, based on a patients risk score on an electronic medical record HIV prediction model, referrals from providers and/or patient self-referrals, a PrEP patient navigator will meet with individuals at the jail to discuss HIV risk, offer HIV/STI testing if not yet completed and offer education around PrEP with referrals to community-based PrEP providers.

DETAILED DESCRIPTION:
The objective of Aim 3 is to deploy the multicomponent strategy that was refined in Aim 2 and evaluate its impact on PrEP implementation and related clinical outcomes using iterative quantitative and qualitative assessments. The investigators' approach will be to utilize the EPIS framework (Exploration, Preparation, Implementation, Sustainment) across the jail-to-community continuum. The investigators will use mixed-methods to evaluate implementation process measures and an interrupted time series design to measure clinical outcomes for PrEP evaluations and linkage, as well as HIV/STI testing and diagnoses. The investigators' expected outcome is to define a feasible, acceptable and effective PrEP implementation strategy for jails.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Incarcerated in Dallas County Jail

Exclusion Criteria:

* Severe medical or psychiatric disability making participation unsafe
* Unable to provide consent
* Not remaining in the local area after release from custody

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Linkage to PrEP care | Within 90 days of release from jail
  Measure the proportion of individuals (of those who stated that they were interested in PrEP and have been released from jail) who attended a clinic visit with a PrEP provider as confirmed by the PrEP patient navigator or through medical record review.

CONTACTS AND LOCATIONS:
Overall Officials: Ank Nijhawan, MD, Principal Investigator — University of Texas Southwestern Medical Center; Douglas Krakower, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Dallas County Jail, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
MPIs will consider de-identified data sharing upon reasonable request from other researchers